CLINICAL TRIAL: NCT00951717
Title: Preparation and Patient Education to Reduce Postpartum Depressive Symptoms
Brief Title: Using a Preparation and Education Intervention to Reduce Postpartum Depression Among New Mothers (The MADE IT 2 Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05-1062; R01MH077683 (NIH); DSIR 83-ATP
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Depression, Postpartum; Depression
Keywords: Postpartum Depressive Symptoms; Physical Symptoms; Emotional Symptoms; Infant Colic; Social Support; Breastfeeding
MeSH Terms: conditions — Depression, Postpartum; Depression; Colic; Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual (No Intervention): Participants will receive standard postpartum education and discharge materials provided by the hospital and a list of community and Internet resources by mail.
- Behavioral education (Experimental): Participants will receive behavioral education on postpartum depression and a list of community and Internet resources by mail.
  Interventions: Behavioral: Behavioral education intervention

INTERVENTIONS:
Behavioral: Behavioral education intervention — One education session with a social worker while at the hospital, provision of an educational pamphlet and summary sheet for partner, a needs assessment by the social worker 2 weeks after hospital discharge, and additional patient education and reinforcement of self-management skills, as needed
  Arms: Behavioral education

SUMMARY:
This study will test an intervention that aims to prevent postpartum depression by providing new mothers with information on and resources for dealing with the disorder.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a disorder affecting many women after delivery of a child. Up to 50% of mothers may experience some depressive symptoms after giving birth, and up to 25% of them will develop major depressive disorder. Some situational factors that place mothers at risk of PPD may be changed or minimized, including social support, the mother's efficiency in handling situational stress, and distress from physical symptoms. Preparing mothers to identify potential situational triggers of depressive symptoms, enhancing their postpartum self-management skills, and providing them access to the proper social and healthcare resources may prevent them from developing major depression. This study will test the efficacy of a brief intervention that aims to prevent PPD by preparing mothers to deal with stressful triggers and depressive symptoms.

This study will last 6 months. Participants will be randomly assigned to receive either treatment as usual or the behavioral education intervention. The intervention will involve two parts. First, after giving birth and while still in the hospital, participants will complete an education session with a social worker and receive written materials about PPD. Then, 2 weeks after discharge from the hospital, participants will receive a call from the social worker, who will conduct a needs assessment that addresses participants' physical and emotional health. If a participant is experiencing distress, the social worker will refer her to appropriate resources and will reinforce self-management skills. All participants will receive a list of community and hospital resources by mail.

Study assessments will take place at 3 weeks, 3 months, and 6 months after study entry. At these points, participants will complete a 20-minute phone survey with a research assistant about their health, mood, and basic demographic information.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the Maternity Unit at Mount Sinai Hospital
* Infant has a birth weight greater than or equal to 2,500 grams
* Infant has a 5-minute Apgar score greater than or equal to 7
* Self-identifies as White or minority other than Black or Hispanic; Black and Hispanic women will be referred to a parallel study with the same protocol at Mount Sinai Hospital
* Speaks English
* Has a working telephone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Measured at baseline
Depressive symptoms | Measured at 3 weeks
Depressive symptoms | Measured at 3 months
Depressive symptoms | Measured at 6 months

SECONDARY OUTCOMES:
Breastfeeding continuation rate | Measured at baseline
Breastfeeding continuation rate | Measured at 3 weeks
Breastfeeding continuation rate | Measured at 3 months
Breastfeeding continuation rate | Measured at 6 months
Physical functioning | Measured at baseline
Physical functioning | Measured at 3 weeks
Physical functioning | Measured at 3 months
Physical functioning | Measured at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Howell, MD, MPP, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

REFERENCES:
- [Derived] Bodnar-Deren S, Klipstein K, Fersh M, Shemesh E, Howell EA. Suicidal Ideation During the Postpartum Period. J Womens Health (Larchmt). 2016 Dec;25(12):1219-1224. doi: 10.1089/jwh.2015.5346. Epub 2016 May 26. PMID 27227751
- [Derived] Balbierz A, Bodnar-Deren S, Wang JJ, Howell EA. Maternal depressive symptoms and parenting practices 3-months postpartum. Matern Child Health J. 2015 Jun;19(6):1212-9. doi: 10.1007/s10995-014-1625-6. PMID 25374288
- [Derived] Howell EA, Bodnar-Deren S, Balbierz A, Loudon H, Mora PA, Zlotnick C, Wang J, Leventhal H. An intervention to reduce postpartum depressive symptoms: a randomized controlled trial. Arch Womens Ment Health. 2014 Feb;17(1):57-63. doi: 10.1007/s00737-013-0381-8. Epub 2013 Sep 10. PMID 24019052
- [Derived] Negron R, Martin A, Almog M, Balbierz A, Howell EA. Social support during the postpartum period: mothers' views on needs, expectations, and mobilization of support. Matern Child Health J. 2013 May;17(4):616-23. doi: 10.1007/s10995-012-1037-4. PMID 22581378